CLINICAL TRIAL: NCT01454102
Title: A Multi-arm Phase I Safety Study of Nivolumab in Combination With Gemcitabine/Cisplatin, Pemetrexed/Cisplatin, Carboplatin/Paclitaxel, Bevacizumab Maintenance, Erlotinib, Ipilimumab or as Monotherapy in Subjects With Stage IIIB/IV Non-small Cell Lung Cancer (NSCLC)
Brief Title: Study of Nivolumab (BMS-936558) in Combination With Gemcitabine/Cisplatin, Pemetrexed/Cisplatin, Carboplatin/Paclitaxel, Bevacizumab Maintenance, Erlotinib, Ipilimumab or as Monotherapy in Subjects With Stage IIIB/IV Non-small Cell Lung Cancer (NSCLC) (CheckMate 012)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-012
Record Dates: First submitted 2011-09-16; First posted 2011-10-18 (Estimated); Results first posted 2019-08-05 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-09

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab; Gemcitabine; Cisplatin; Pemetrexed; Paclitaxel; Carboplatin; Bevacizumab; Erlotinib Hydrochloride; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (19):
- Arm A: Nivolumab + Gemcitabine + Cisplatin (Experimental): Nivolumab solution intravenously every 3 weeks until progressive disease (PD) or discontinuation due to toxicity. Administered prior to chemotherapy on Day 1 of each cycle
  Gemcitabine solution intravenously on Day 1 and Day 8 of every cycle for 4 cycles
  Cisplatin solution intravenously on Day 1 of each cycle for 4 cycles
  Interventions: Biological: Nivolumab; Drug: Gemcitabine; Drug: Cisplatin
- Arm B: Nivolumab + Pemetrexed + Cisplatin (Experimental): Nivolumab solution intravenously every 3 weeks until PD or discontinuation due to toxicity. Administered prior to chemotherapy on Day 1 of each cycle
  Pemetrexed solution intravenously on Day 1 of every cycle for 4 cycles
  Cisplatin solution intravenously on Day 1 of each cycle for 4 cycles
  Interventions: Biological: Nivolumab; Drug: Cisplatin; Drug: Pemetrexed
- Arm C: Nivolumab + Paclitaxel + Carboplatin (Experimental): Nivolumab solution intravenously every 3 weeks until PD or discontinuation due to toxicity. Administered prior to chemotherapy on Day 1 of each cycle
  Paclitaxel solution intravenously on Day 1 of every cycle for 4 cycles
  Carboplatin area under curve (AUC) 6 solution intravenously on Day 1 of every cycle for 4 cycles
  Interventions: Biological: Nivolumab; Drug: Paclitaxel; Drug: Carboplatin
- Arm D: Nivolumab + Bevacizumab maintenance (Experimental): Nivolumab solution intravenously every 3 weeks until PD or discontinuation due to toxicity. Administered prior to chemotherapy on Day 1 of each cycle
  Bevacizumab administered prior to intravenous infusion on Cycle 1 Day 1 followed by intravenous infusion every 3 weeks on Cycle 2 onwards and until PD or discontinuation due to toxicity
  Interventions: Biological: Nivolumab; Drug: Bevacizumab
- Arm E: Nivolumab + Erlotinib (Experimental): Nivolumab solution intravenously every 2 weeks until PD or discontinuation due to toxicity. Administered prior to chemotherapy on Day 1 of each cycle
  Erlotinib tablet by mouth daily until PD or discontinuation due to toxicity
  Interventions: Biological: Nivolumab; Drug: Erlotinib
- Arm F: Nivolumab (Experimental): Nivolumab solution intravenously every 2 weeks until PD or discontinuation due to toxicity. Administered over 60 minutes
  Interventions: Biological: Nivolumab
- Arm G: Nivolumab + Ipilimumab (Experimental): In Squamous histology subjects (NSCLC)
  Nivolumab solution administered intravenously prior to Ipilimumab on Day 1 of each cycle. Combination regimen will be provided for 4 cycles
  Ipilimumab solution administered intravenously on Day 1 of each cycle, for 4 cycles
  Followed by Nivolumab administered until PD or discontinuation due to toxicity
  Interventions: Biological: Nivolumab; Biological: Ipilimumab
- Arm H: Nivolumab + Ipilimumab (Experimental): In non-squamous histology subjects (NSCLC)
  Nivolumab solution administered intravenously prior to Ipilimumab on Day 1 of each cycle. Combination regimen will be provided for 4 cycles
  Ipilimumab solution administered intravenously on Day 1 of each cycle, for 4 cycles
  Followed by Nivolumab administered every 2 weeks until PD or discontinuation due to toxicity
  Interventions: Biological: Nivolumab; Biological: Ipilimumab
- Arm I: Nivolumab + Ipilimumab (Experimental): In squamous histology subjects (NSCLC)
  Nivolumab solution administered intravenously prior to Ipilimumab on Day 1 of each cycle. Combination regimen will be provided for 4 cycles
  Ipilimumab solution administered intravenously on Day 1 of each cycle, for 4 cycles
  Followed by Nivolumab administered every 2 weeks until PD or discontinuation due to toxicity
  Interventions: Biological: Nivolumab; Biological: Ipilimumab
- Arm J: Nivolumab + Ipilimumab (Experimental): In non-squamous histology subjects (NSCLC)
  Nivolumab solution administered intravenously prior to Ipilimumab on Day 1 of each cycle. Combination regimen will be provided for 4 cycles
  Ipilimumab solution administered intravenously on Day 1 of each cycle, for 4 cycles
  Followed by Nivolumab administered every 2 weeks until PD or discontinuation due to toxicity
  Interventions: Biological: Nivolumab; Biological: Ipilimumab
- Arm K: Nivolumab (Experimental): In squamous histology subjects (NSCLC)
  Nivolumab solution intravenously every 2 weeks until PD or discontinuation due to toxicity. Administered as switch maintenance therapy. A cycle is 2 weeks
  Interventions: Biological: Nivolumab
- Arm L: Nivolumab (Experimental): In non-squamous histology subjects (NSCLC)
  Nivolumab solution intravenously every 2 weeks until PD or discontinuation due to toxicity. Administered over 60 minutes as switch maintenance therapy. A cycle is 2 weeks
  Interventions: Biological: Nivolumab
- Arm M: Nivolumab (Experimental): NSCLC subjects with untreated, asymptomatic brain metastases and have no evidence of cerebral edema
  Nivolumab solution intravenously every 2 weeks until PD or discontinuation due to toxicity. Administered for up to an hour as monotherapy. A cycle is 2 weeks
  Interventions: Biological: Nivolumab
- Arm N: Nivolumab + Ipilimumab (Experimental): In subjects with any histology (NSCLC)
  Nivolumab solution administered intravenously prior to Ipilimumab on Day 1 of each cycle. Combination regimen will be provided for 4 cycles
  Ipilimumab solution administered intravenously on Day 1 of each cycle, for 4 cycles
  Followed by Nivolumab administered every 2 weeks until PD or discontinuation due to toxicity
  Interventions: Biological: Nivolumab; Biological: Ipilimumab
- Arm O: Nivolumab + Ipilimumab (Experimental): Nivolumab at specified dose/schedule until PD or discontinuation due to toxicity
  Ipilimumab at specified dose/schedule until PD or discontinuation due to toxicity
  Interventions: Biological: Nivolumab; Biological: Ipilimumab
- Arm P: Nivolumab + Ipilimumab (Experimental): Nivolumab at specified dose/schedule until PD or discontinuation due to toxicity
  Ipilimumab at specified dose/schedule until PD or discontinuation due to toxicity
  Interventions: Biological: Nivolumab; Biological: Ipilimumab
- Arm Q: Nivolumab + Ipilimumab (Experimental): Nivolumab at specified dose/schedule until PD or discontinuation due to toxicity
  Ipilimumab at specified dose/schedule until PD or discontinuation due to toxicity
  Interventions: Biological: Nivolumab; Biological: Ipilimumab
- Arm R: Nivolumab + Ipilimumab (Experimental): Nivolumab at specified dose/schedule until PD or discontinuation due to toxicity
  Ipilimumab at specified dose/schedule until PD or discontinuation due to toxicity
  Interventions: Biological: Nivolumab; Biological: Ipilimumab
- Arm S: Nivolumab + Ipilimumab (Experimental): Nivolumab at specified dose/schedule until PD or discontinuation due to toxicity
  Ipilimumab at specified dose/schedule until PD or discontinuation due to toxicity
  Interventions: Biological: Nivolumab; Biological: Ipilimumab

INTERVENTIONS:
Biological: Nivolumab
  Other Names: BMS-936558
Drug: Gemcitabine
  Arms: Arm A: Nivolumab + Gemcitabine + Cisplatin
Drug: Cisplatin
  Arms: Arm A: Nivolumab + Gemcitabine + Cisplatin; Arm B: Nivolumab + Pemetrexed + Cisplatin
Drug: Pemetrexed
  Arms: Arm B: Nivolumab + Pemetrexed + Cisplatin
Drug: Paclitaxel
  Arms: Arm C: Nivolumab + Paclitaxel + Carboplatin
Drug: Carboplatin
  Arms: Arm C: Nivolumab + Paclitaxel + Carboplatin
Drug: Bevacizumab
  Arms: Arm D: Nivolumab + Bevacizumab maintenance
Drug: Erlotinib
  Arms: Arm E: Nivolumab + Erlotinib
Biological: Ipilimumab
  Arms: Arm G: Nivolumab + Ipilimumab; Arm H: Nivolumab + Ipilimumab; Arm I: Nivolumab + Ipilimumab; Arm J: Nivolumab + Ipilimumab; Arm N: Nivolumab + Ipilimumab; Arm O: Nivolumab + Ipilimumab; Arm P: Nivolumab + Ipilimumab; Arm Q: Nivolumab + Ipilimumab; Arm R: Nivolumab + Ipilimumab; Arm S: Nivolumab + Ipilimumab

SUMMARY:
* The study is evaluating the safety and tolerability of Nivolumab (BMS-936558) when combined with three platinum-based doublet chemotherapy regimens (Cisplatin/Gemcitabine; Cisplatin/Pemetrexed; and Carboplatin/Paclitaxel) in subjects with NSCLC.
* The study is evaluating the safety and tolerability of Nivolumab as maintenance therapy in combination with Bevacizumab/Avastin that will be given after at least 4 cycles of platinum doublet chemotherapy.
* The study is evaluating the safety and tolerability of Nivolumab in combination with Erlotinib among epidermal growth factor receptor (EGFR) mutation positive non-squamous NSCLC subjects and as monotherapy in subjects with NSCLC.
* The study is evaluating the safety and tolerability of Nivolumab in combination with Ipilimumab in subjects with squamous and non-squamous NSCLC.
* The study is evaluating the safety and tolerability of Nivolumab as switch maintenance therapy in subjects with squamous and non-squamous NSCLC.
* The study is evaluating the safety and tolerability of Nivolumab as monotherapy among subjects with untreated, asymptomatic brain metastases and no evidence of cerebral edema.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Newly diagnosed and confirmed Stage IIIB/IV NSCLC
* Previously treated NSCLC with asymptomatic brain metastases (eligible for Arm M) See additional details below
* Men and women aged ≥18 years
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* Subject must be chemotherapy naive (except Arm D, K, L and M). Prior use of epidermal growth factor receptor (EGFR) tyrosine kinase inhibitor (TKI) is acceptable. For Arms D, K, and L, subjects must be non-progressors within 42 days after completion of first-line treatment with ≥4 cycles of Platinum Doublet chemotherapy with or without Bevacizumab. See below for Arm M
* Either a formalin fixed tissue block or a minimum of 10 slides of tumor sample (archived or fresh) must be available for biomarker evaluation (a local pathologist must review for adequacy of sampling)
* Life expectancy of at least 3 months
* Prior radiotherapy must have been completed at least 2 weeks prior to study entry

For Arm M:

* No more than 4 brain metastases
* Each brain metastases ≤3 cm in size
* No evidence of cerebral edema
* Subjects must be free of neurologic symptoms related to metastatic brain lesions and must not have required or received systemic corticosteroids for ≥10 days prior to initiation of study treatment
* At least 1 measurable target brain lesion >0.5 cm and no larger than 3 cm in diameter and/or 2 measurable brain target lesions >0.3 cm
* No prior radiation therapy, surgery, or other local therapy for target brain lesions
* Must have received at least one prior systemic anticancer therapy for NSCLC

Exclusion Criteria:

* Subjects with symptomatic brain metastases, spinal cord compression, or intractable back pain due to a compressive or destructive mass
* Subjects who require emergent use of systemic steroids, emergent surgery and/or radiotherapy
* Any active or history of a known autoimmune disease
* Subjects with previous malignancies (except non-melanoma skin cancers, in situ bladder cancer, gastric, or colon cancers or cervical cancers/dysplasia, or breast carcinoma in situ) are excluded unless a complete remission was achieved at least 2 years prior to study entry and no additional therapy is required or anticipated to be required during the study period
* History of Grade ≥2 neuropathy
* Subjects with interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 472 (Actual)
Dates: Start 2011-12-16 (Actual); Primary Completion 2016-07-20 (Actual); Study Completion 2021-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (12):
- United States (9):
  - Ucla, Los Angeles, California
  - Yale University, New Haven, Connecticut
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Memorial Sloan Kettering Nassau, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Ut Southwestern Medical Center At Dallas, Dallas, Texas
  - University of Washington - Seattle Cancer Care Alliance, Seattle, Washington
- Canada (3):
  - Local Institution, Hamilton, Ontario
  - Local Institution, Ottawa, Ontario
  - Local Institution, Toronto, Ontario

REFERENCES:
- [Background] Gettinger S, Rizvi NA, Chow LQ, Borghaei H, Brahmer J, Ready N, Gerber DE, Shepherd FA, Antonia S, Goldman JW, Juergens RA, Laurie SA, Nathan FE, Shen Y, Harbison CT, Hellmann MD. Nivolumab Monotherapy for First-Line Treatment of Advanced Non-Small-Cell Lung Cancer. J Clin Oncol. 2016 Sep 1;34(25):2980-7. doi: 10.1200/JCO.2016.66.9929. Epub 2016 Jun 27. PMID 27354485
- [Background] Rizvi NA, Hellmann MD, Brahmer JR, Juergens RA, Borghaei H, Gettinger S, Chow LQ, Gerber DE, Laurie SA, Goldman JW, Shepherd FA, Chen AC, Shen Y, Nathan FE, Harbison CT, Antonia S. Nivolumab in Combination With Platinum-Based Doublet Chemotherapy for First-Line Treatment of Advanced Non-Small-Cell Lung Cancer. J Clin Oncol. 2016 Sep 1;34(25):2969-79. doi: 10.1200/JCO.2016.66.9861. Epub 2016 Jun 27. PMID 27354481
- [Background] Hellmann MD, Rizvi NA, Goldman JW, Gettinger SN, Borghaei H, Brahmer JR, Ready NE, Gerber DE, Chow LQ, Juergens RA, Shepherd FA, Laurie SA, Geese WJ, Agrawal S, Young TC, Li X, Antonia SJ. Nivolumab plus ipilimumab as first-line treatment for advanced non-small-cell lung cancer (CheckMate 012): results of an open-label, phase 1, multicohort study. Lancet Oncol. 2017 Jan;18(1):31-41. doi: 10.1016/S1470-2045(16)30624-6. Epub 2016 Dec 5. PMID 27932067
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 472 participants were enrolled; 376 participants received at least one dose of study treatment
Groups:
- Arm A: Nivolumab + Gemcitabine + Cisplatin: Chemotherapy-naive SQ subjects; GEM 1250 mg/m2 Days 1 and 8 with CIS 75 mg/m2 on Day 1 of a Q3W cycle for up to 4 cycles + Nivo 10 mg/kg Q3W until progression after cycle 4
- Arm B: Nivolumab + Pemetrexed + Cisplatin: Chemotherapy-naive NSQ subjects; dose de-escalation design; PEM 500 mg/m2 with CIS 75 mg/m2, both on Day 1 of a Q3W cycle for up to 4 cycles + Nivo 10 mg/kg Q3W until progression after cycle 4
- Arm C10: Nivolumab + Paclitaxel + Carboplatin: Chemotherapy-naive subjects with any histology; dose de-escalation design; PAC 200 mg/m2 with CAR AUC 6, both on Day 1 of a Q3W cycle for up to 4 cycles + Nivo 10 mg/kg Q3W until progression after cycle 4
- Arm D: Nivolumab + Bevacizumab Maintenance: NSQ subjects who completed >= 4 cycles of chemotherapy and are nonprogressors; BEV 15 mg/kg + Nivo 5 mg/kg Q3W until progression
- Arm E: Nivolumab + Erlotinib: Chemotherapy-naive, subjects with EGFR mutations; ERL 150 mg PO, daily + Nivo 3 mg/kg Q2W until progression
- Arm F: Nivolumab: Chemotherapy-naive subjects with any histology; Nivo 3 mg/kg Q2W until progression
- Arm GH: Nivolumab + Ipilimumab: Chemotherapy-naive SQ and NSQ subjects; Nivo 1 mg/kg + Ipi 3 mg/kg Q3W for 4 cycles followed by Nivo 3 mg/kg Q2W until progression
- Arm IJ: Nivolumab + Ipilimumab: Chemotherapy-naive SQ and NSQ subjects; Nivo 3 mg/kg + Ipi 1 mg/kg Q3W for 4 cycles followed by Nivo 3 mg/kg Q2W until progression
- Arm K: Nivolumab in Squamous Histology Subjects (NSCLC): SQ subjects who completed >= 4 cycles of chemotherapy and are nonprogressors; Nivo 3 mg/kg Q2W as switch maintenance therapy until progression
- Arm L: Nivolumab in Non-squamous Histology Subjects (NSCLC): NSQ subjects who completed >= 4 cycles of chemotherapy and are nonprogressors; Nivo 3 mg/kg Q2W as switch maintenance therapy until progression
- Arm M: Nivolumab: Subjects with any histology and untreated, asymptomatic brain metastases; Nivo 3 mg/kg Q2W until progression
- Arm N: Nivolumab + Ipilimumab: Chemotherapy-naive subjects with any histology; Nivo 1 mg/kg + Ipi 1 mg/kg Q3W for 4 cycles followed by Nivo 3 mg/kg Q2W until progression
- Arm O: Nivolumab + Ipilimumab: Chemotherapy-naive subjects with any histology; Nivo 1 mg/kg Q2W + Ipi 1 mg/kg Q6W until progression or unacceptable toxicity
- Arm P: Nivolumab + Ipilimumab: Chemotherapy-naive subjects with any histology; Nivo 3 mg/kg Q2W + Ipi 1 mg/kg Q12W until progression or unacceptable toxicity
- Arm Q: Nivolumab + Ipilimumab: Chemotherapy-naive subjects with any histology; Nivo 3 mg/kg Q2W + Ipi 1 mg/kg Q6W until progression or unacceptable toxicity
- Arm C5: Nivolumab + Paclitaxel + Carboplatin: Chemotherapy-naive subjects with any histology; dose de-escalation design; PAC 200 mg/m2 with CAR AUC 6, both on Day 1 of a Q3W cycle for up to 4 cycles + Nivo 5 mg/kg Q3W until progression after cycle 4
Period: Overall Study
Arm/Group | Arm A: Nivolumab + Gemcitabine + Cisplatin | Arm B: Nivolumab + Pemetrexed + Cisplatin | Arm C10: Nivolumab + Paclitaxel + Carboplatin | Arm D: Nivolumab + Bevacizumab Maintenance | Arm E: Nivolumab + Erlotinib | Arm F: Nivolumab | Arm GH: Nivolumab + Ipilimumab | Arm IJ: Nivolumab + Ipilimumab | Arm K: Nivolumab in Squamous Histology Subjects (NSCLC) | Arm L: Nivolumab in Non-squamous Histology Subjects (NSCLC) | Arm M: Nivolumab | Arm N: Nivolumab + Ipilimumab | Arm O: Nivolumab + Ipilimumab | Arm P: Nivolumab + Ipilimumab | Arm Q: Nivolumab + Ipilimumab | Arm C5: Nivolumab + Paclitaxel + Carboplatin
Started | 12 | 15 | 15 | 12 | 21 | 52 | 24 | 25 | 13 | 13 | 12 | 31 | 40 | 38 | 39 | 14
Completed | 12 | 15 | 15 | 12 | 18 | 49 | 22 | 25 | 12 | 13 | 12 | 27 | 33 | 34 | 36 | 13
Not Completed | 0 | 0 | 0 | 0 | 3 | 3 | 2 | 0 | 1 | 0 | 0 | 4 | 7 | 4 | 3 | 1
Not completed — Continuing in the treatment period | 0 | 0 | 0 | 0 | 3 | 3 | 2 | 0 | 1 | 0 | 0 | 4 | 7 | 4 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Nivolumab + Gemcitabine + Cisplatin | Arm B: Nivolumab + Pemetrexed + Cisplatin | Arm C10: Nivolumab + Paclitaxel + Carboplatin | Arm D: Nivolumab + Bevacizumab Maintenance | Arm E: Nivolumab + Erlotinib | Arm F: Nivolumab | Arm GH: Nivolumab + Ipilimumab | Arm IJ: Nivolumab + Ipilimumab | Arm K: Nivolumab in Squamous Histology Subjects (NSCLC) | Arm L: Nivolumab in Non-squamous Histology Subjects (NSCLC) | Arm M: Nivolumab | Arm N: Nivolumab + Ipilimumab | Arm O: Nivolumab + Ipilimumab | Arm P: Nivolumab + Ipilimumab | Arm Q: Nivolumab + Ipilimumab | Arm C5: Nivolumab + Paclitaxel + Carboplatin | Total
Number analyzed (Participants) | 12 | 15 | 15 | 12 | 21 | 52 | 24 | 25 | 13 | 13 | 12 | 31 | 40 | 38 | 39 | 14 | 376
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (6.82) | 60.2 (11.20) | 58.7 (8.81) | 62.9 (9.53) | 62.8 (9.41) | 67.0 (9.96) | 60.5 (6.99) | 63.1 (8.31) | 63.6 (10.15) | 68.7 (12.64) | 62.6 (12.65) | 61.5 (10.85) | 64.9 (11.25) | 65.9 (9.36) | 64.4 (9.95) | 64.9 (9.79) | 64.0 (9.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 8 | 5 | 13 | 26 | 10 | 12 | 5 | 5 | 8 | 16 | 22 | 21 | 15 | 8 | 188
  Male | 7 | 6 | 7 | 7 | 8 | 26 | 14 | 13 | 8 | 8 | 4 | 15 | 18 | 17 | 24 | 6 | 188

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Serious Adverse Events (SAE), Adverse Events (AE) Leading to Discontinuation, or Death
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Treatment-related=having certain, probable, possible, or missing relationship to study drug. Grade (Gr) 1=Mild, Gr 2=Moderate, Gr 3=Severe, Gr 4= Potentially Life-threatening or disabling.
Time Frame: From first dose to 30 days after the last dose of study drug (assessed up to July 2016, approximately 55 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Nivolumab + Gemcitabine + Cisplatin | Arm B: Nivolumab + Pemetrexed + Cisplatin | Arm C10: Nivolumab + Paclitaxel + Carboplatin | Arm D: Nivolumab + Bevacizumab Maintenance | Arm E: Nivolumab + Erlotinib | Arm F: Nivolumab | Arm GH: Nivolumab + Ipilimumab | Arm IJ: Nivolumab + Ipilimumab | Arm K: Nivolumab in Squamous Histology Subjects (NSCLC) | Arm L: Nivolumab in Non-squamous Histology Subjects (NSCLC) | Arm M: Nivolumab | Arm N: Nivolumab + Ipilimumab | Arm O: Nivolumab + Ipilimumab | Arm P: Nivolumab + Ipilimumab | Arm Q: Nivolumab + Ipilimumab | Arm C5: Nivolumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 12 | 15 | 15 | 12 | 21 | 52 | 24 | 25 | 13 | 13 | 12 | 31 | 40 | 38 | 39 | 14
Participants
  SAEs | 4 | 10 | 8 | 3 | 11 | 23 | 18 | 17 | 3 | 4 | 4 | 12 | 21 | 25 | 25 | 9
  AEs leading to discontinuation | 2 | 5 | 1 | 3 | 3 | 9 | 11 | 13 | 3 | 4 | 1 | 3 | 4 | 10 | 8 | 2
  Death | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 3 | 0 | 1 | 1 | 1 | 1 | 4 | 2 | 0

2. Primary Outcome: Number of Participants Who Experienced Selected Adverse Events
Description: The number of participants who experienced an AE of interest due to any cause is presented. Endocrine, Gastrointestinal, Hepatic, Pulmonary, Renal, Skin, and
  Hypersensitivity/Infusion select AEs were identified that are potentially associated with the use of nivolumab, based on the following 4 guiding principles:
  * AEs that may differ in type, frequency, or severity from AEs caused by non-immunotherapies
  * AEs that may require immunosuppression (eg, corticosteroids) as part of their management
  * AEs whose early recognition and management may mitigate severe toxicity
  * AEs for which multiple event terms may be used to describe a single type of AE, thereby necessitating the pooling of terms for full characterization.
Time Frame: From first dose to 30 days after the last dose of study drug (assessed up to July 2016, approximately 55 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Nivolumab + Gemcitabine + Cisplatin | Arm B: Nivolumab + Pemetrexed + Cisplatin | Arm C10: Nivolumab + Paclitaxel + Carboplatin | Arm D: Nivolumab + Bevacizumab Maintenance | Arm E: Nivolumab + Erlotinib | Arm F: Nivolumab | Arm GH: Nivolumab + Ipilimumab | Arm IJ: Nivolumab + Ipilimumab | Arm K: Nivolumab in Squamous Histology Subjects (NSCLC) | Arm L: Nivolumab in Non-squamous Histology Subjects (NSCLC) | Arm M: Nivolumab | Arm N: Nivolumab + Ipilimumab | Arm O: Nivolumab + Ipilimumab | Arm P: Nivolumab + Ipilimumab | Arm Q: Nivolumab + Ipilimumab | Arm C5: Nivolumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 12 | 15 | 15 | 12 | 21 | 52 | 24 | 25 | 13 | 13 | 12 | 31 | 40 | 38 | 39 | 14
Participants
  Endorcrine | 3 | 2 | 0 | 2 | 4 | 8 | 8 | 6 | 3 | 2 | 0 | 4 | 15 | 8 | 12 | 1
  Gastrointestinal | 4 | 6 | 8 | 2 | 10 | 16 | 15 | 12 | 5 | 1 | 1 | 12 | 13 | 11 | 13 | 6
  Hepatic | 0 | 2 | 1 | 0 | 4 | 5 | 7 | 2 | 2 | 0 | 0 | 4 | 13 | 1 | 2 | 0
  Pulmonary | 2 | 2 | 0 | 2 | 1 | 3 | 3 | 2 | 1 | 2 | 0 | 3 | 3 | 5 | 3 | 1
  Renal | 1 | 6 | 1 | 1 | 2 | 0 | 2 | 0 | 3 | 0 | 0 | 2 | 2 | 6 | 4 | 4
  Skin | 3 | 9 | 7 | 5 | 16 | 27 | 15 | 14 | 4 | 2 | 2 | 20 | 20 | 21 | 20 | 7
  Hypersensitivity/Infusion Reactions | 1 | 6 | 7 | 1 | 2 | 4 | 1 | 3 | 2 | 0 | 0 | 1 | 1 | 3 | 1 | 1

3. Primary Outcome: Number of Participants With Abnormalities in Selected Hepatic Clinical Laboratory Tests
Description: The number of subjects with selected hepatic laboratory abnormalities is reported.
  AST= aspartate aminotransferase; ALT= alanine aminotransferase; ULN= upper limit of normal.
Time Frame: From first dose to 30 days following last dose of study drug (assessed up to July 2016, approximately 55 months)
Population: All treated participants with baseline and post-baseline measurements
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Nivolumab + Gemcitabine + Cisplatin | Arm B: Nivolumab + Pemetrexed + Cisplatin | Arm C10: Nivolumab + Paclitaxel + Carboplatin | Arm D: Nivolumab + Bevacizumab Maintenance | Arm E: Nivolumab + Erlotinib | Arm F: Nivolumab | Arm GH: Nivolumab + Ipilimumab | Arm IJ: Nivolumab + Ipilimumab | Arm K: Nivolumab in Squamous Histology Subjects (NSCLC) | Arm L: Nivolumab in Non-squamous Histology Subjects (NSCLC) | Arm M: Nivolumab | Arm N: Nivolumab + Ipilimumab | Arm O: Nivolumab + Ipilimumab | Arm P: Nivolumab + Ipilimumab | Arm Q: Nivolumab + Ipilimumab | Arm C5: Nivolumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 12 | 15 | 14 | 12 | 20 | 51 | 24 | 24 | 12 | 13 | 11 | 29 | 37 | 37 | 36 | 14
Participants
  ALT OR AST > 3XULN | 0 | 0 | 2 | 1 | 4 | 2 | 6 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 2
  ALT OR AST > 5XULN | 0 | 0 | 0 | 0 | 2 | 2 | 4 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  ALT OR AST > 10XULN | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  ALT OR AST > 20XULN | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  TOTAL BILIRUBIN > 2XULN | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST or ALT>3XULN with Bilirubin>2XULN within 1 day | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST or ALT>3XULN with Bilirubin>2XULN within 30day | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Abnormalities in Selected Thyroid Clinical Laboratory Tests
Description: The number of subjects with selected thyroid laboratory abnormalities is reported. FT3 and FT4 test abnormalities were considered for a 2-week window after the abnormal TSH test date.
  TSH= thyroid-stimulating hormone; FT3= Free T3; FT4= Free T4; LLN= lower limit of normal; ULN= upper limit of normal
Time Frame: From first dose to 30 days following last dose of study drug (assessed up to July 2016, approximately 55 months)
Population: All treated participants with baseline and post-baseline measurements
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Nivolumab + Gemcitabine + Cisplatin | Arm B: Nivolumab + Pemetrexed + Cisplatin | Arm C10: Nivolumab + Paclitaxel + Carboplatin | Arm D: Nivolumab + Bevacizumab Maintenance | Arm E: Nivolumab + Erlotinib | Arm F: Nivolumab | Arm GH: Nivolumab + Ipilimumab | Arm IJ: Nivolumab + Ipilimumab | Arm K: Nivolumab in Squamous Histology Subjects (NSCLC) | Arm L: Nivolumab in Non-squamous Histology Subjects (NSCLC) | Arm M: Nivolumab | Arm N: Nivolumab + Ipilimumab | Arm O: Nivolumab + Ipilimumab | Arm P: Nivolumab + Ipilimumab | Arm Q: Nivolumab + Ipilimumab | Arm C5: Nivolumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 12 | 14 | 14 | 12 | 20 | 51 | 23 | 23 | 12 | 13 | 11 | 29 | 34 | 34 | 28 | 14
Participants
  TSH > ULN | 2 | 3 | 1 | 8 | 12 | 21 | 10 | 7 | 5 | 5 | 2 | 10 | 12 | 11 | 11 | 5
  TSH > ULN WITH TSH <= ULN AT BASELINE | 1 | 2 | 1 | 4 | 8 | 13 | 10 | 6 | 5 | 3 | 1 | 7 | 9 | 5 | 8 | 4
  TSH > ULN WITH >=1 FT3/FT4 TEST VALUE < LLN | 0 | 1 | 0 | 1 | 7 | 3 | 5 | 5 | 3 | 0 | 0 | 6 | 7 | 5 | 4 | 2
  TSH > ULN WITH ALL FT3/FT4 TEST VALUES >= LLN | 0 | 2 | 1 | 0 | 0 | 4 | 1 | 2 | 2 | 2 | 0 | 1 | 1 | 0 | 2 | 0
  TSH > ULN WITH FT3/FT4 TEST MISSING | 2 | 0 | 0 | 7 | 5 | 14 | 4 | 0 | 0 | 3 | 2 | 3 | 4 | 6 | 5 | 3
  TSH < LLN | 2 | 7 | 5 | 2 | 7 | 9 | 12 | 9 | 3 | 1 | 6 | 9 | 10 | 6 | 9 | 7
  TSH < LLN WITH TSH >= LLN AT BASELINE | 1 | 3 | 1 | 1 | 7 | 9 | 12 | 9 | 3 | 0 | 4 | 9 | 9 | 6 | 9 | 5
  TSH < LLN WITH >=1 FT3/FT4 TEST VALUE > ULN | 1 | 1 | 0 | 0 | 4 | 4 | 6 | 5 | 2 | 1 | 1 | 6 | 7 | 1 | 1 | 2
  TSH < LLN WITH ALL FT3/FT4 TEST VALUES <= ULN | 0 | 3 | 1 | 1 | 0 | 1 | 3 | 1 | 1 | 0 | 0 | 2 | 2 | 1 | 1 | 0
  TSH < LLN WITH FT3/FT4 TEST MISSING | 1 | 3 | 4 | 1 | 3 | 4 | 3 | 3 | 0 | 0 | 5 | 1 | 1 | 4 | 7 | 5

5. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of all treated participants who achieved a Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR) using the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria as per investigator assessment. This proportion was multiplied by 100 and expressed as a percentage. BOR was defined as the best response designation recorded between the date of randomization and the date of progression, or the date of subsequent anticancer therapy, whichever occurred first. CR or PR determinations included in the BOR assessment were confirmed by a second scan at least 4 weeks after the criteria for responses were first met. For participants without progression or subsequent therapy, all available response designations contributed to the BOR determination. For participants who continued treatment beyond progression, the BOR was determined based on response designations recorded up to the time of the initial progression.
Time Frame: From first dose until date of progression or subsequent anti-cancer therapy (assessed up to July 2016, approximately 55 months)
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Nivolumab + Gemcitabine + Cisplatin | Arm B: Nivolumab + Pemetrexed + Cisplatin | Arm C10: Nivolumab + Paclitaxel + Carboplatin | Arm D: Nivolumab + Bevacizumab Maintenance | Arm E: Nivolumab + Erlotinib | Arm F: Nivolumab | Arm GH: Nivolumab + Ipilimumab | Arm IJ: Nivolumab + Ipilimumab | Arm K: Nivolumab in Squamous Histology Subjects (NSCLC) | Arm L: Nivolumab in Non-squamous Histology Subjects (NSCLC) | Arm M: Nivolumab | Arm N: Nivolumab + Ipilimumab | Arm O: Nivolumab + Ipilimumab | Arm P: Nivolumab + Ipilimumab | Arm Q: Nivolumab + Ipilimumab | Arm C5: Nivolumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 12 | 15 | 15 | 12 | 21 | 52 | 24 | 25 | 13 | 13 | 12 | 31 | 40 | 38 | 39 | 14
Percentage of participants | 41.7 [15.2 to 72.3] | 46.7 [21.3 to 73.4] | 46.7 [21.3 to 73.4] | 16.7 [2.1 to 48.4] | 19.0 [5.4 to 41.9] | 23.1 [12.5 to 36.8] | 20.8 [7.1 to 42.2] | 24.0 [9.4 to 45.1] | 0 [0.0 to 24.7] | 15.4 [1.9 to 45.4] | 8.3 [0.2 to 38.5] | 22.6 [9.6 to 41.1] | 32.5 [18.6 to 49.1] | 47.4 [31.0 to 64.2] | 38.5 [23.4 to 55.4] | 50.0 [23.0 to 77.0]

6. Secondary Outcome: Progression-Free Survival Rate (PFSR) at Week 24
Description: Progression-Free Survival (PFS) was defined as the time from the date of first dose of study medication to the date of first disease progression or death, if death occurred within 100 days of the final dose of study drug. Among participants without previous RECIST-defined progression, participants who died beyond 100 days and those who remained alive were censored at the last tumor assessment date (before subsequent therapy).
  PFSR at week 24 was defined as the proportion of subjects remaining progression free and surviving at 24 weeks. The proportion was calculated by the product-limit method (Kaplan-Meier estimate), which takes into account censored data, and expressed as a percentage.
Time Frame: 24 weeks
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Nivolumab + Gemcitabine + Cisplatin | Arm B: Nivolumab + Pemetrexed + Cisplatin | Arm C10: Nivolumab + Paclitaxel + Carboplatin | Arm D: Nivolumab + Bevacizumab Maintenance | Arm E: Nivolumab + Erlotinib | Arm F: Nivolumab | Arm GH: Nivolumab + Ipilimumab | Arm IJ: Nivolumab + Ipilimumab | Arm K: Nivolumab in Squamous Histology Subjects (NSCLC) | Arm L: Nivolumab in Non-squamous Histology Subjects (NSCLC) | Arm M: Nivolumab | Arm N: Nivolumab + Ipilimumab | Arm O: Nivolumab + Ipilimumab | Arm P: Nivolumab + Ipilimumab | Arm Q: Nivolumab + Ipilimumab | Arm C5: Nivolumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 12 | 15 | 15 | 12 | 21 | 52 | 24 | 25 | 13 | 13 | 12 | 31 | 40 | 38 | 39 | 14
Percentage of participants | 50.5 [18.7 to 75.7] | 68.4 [35.9 to 86.8] | 34.3 [11.3 to 59.2] | 58.3 [27.0 to 80.1] | 50.6 [27.7 to 69.7] | 39.7 [26.0 to 53.1] | 42.8 [22.4 to 61.8] | 37.3 [18.1 to 56.7] | 50.0 [20.8 to 73.6] | 20.5 [3.3 to 47.8] | 8.3 [0.5 to 31.1] | 49.1 [30.3 to 65.5] | 48.0 [31.6 to 62.7] | 72.4 [54.7 to 84.1] | 39.5 [24.2 to 54.4] | 59.3 [27.5 to 81.0]

ADVERSE EVENTS:
Time Frame: From first dose to 30 days after the last dose of study drug (assessed up to July 2016, approximately 55 months)
Description: Adverse event data was only collected by cohort and not by dose. All participants in "Arm C10: Nivolumab (10 mg/kg) + Paclitaxel + Carboplatin" and "Arm C5: Nivolumab (5 mg/kg) + Paclitaxel + Carboplatin" were monitored for adverse events under a single "Arm C" as a cohort.
Groups:
- Arm J: Nivolumab + Ipilimumab: Chemotherapy-naive NSQ subjects; Nivo 3 mg/kg + Ipi 1 mg/kg Q3W for 4 cycles followed by Nivo 3 mg/kg Q2W until progression
- Arm C: Nivolumab + Paclitaxel + Carboplatin: Chemotherapy-naive subjects with any histology; dose de-escalation design; PAC 200 mg/m2 with CAR AUC 6, both on Day 1 of a Q3W cycle for up to 4 cycles + Nivo 10 mg/kg Q3W until progression after cycle 4
- Arm G: Nivolumab + Ipilimumab: Chemotherapy-naive SQ subjects; Nivo 1 mg/kg + Ipi 3 mg/kg Q3W for 4 cycles followed by Nivo 3 mg/kg Q2W until progression
- Arm H: Nivolumab + Ipilimumab: Chemotherapy-naive NSQ subjects; Nivo 1 mg/kg + Ipi 3 mg/kg Q3W for 4 cycles followed by Nivo 3 mg/kg Q2W until progression
- Arm I: Nivolumab + Ipilimumab: Chemotherapy-naive SQ subjects; Nivo 3 mg/kg + Ipi 1 mg/kg Q3W for 4 cycles followed by Nivo 3 mg/kg Q2W until progression
Arm/Group | Arm A: Nivolumab + Gemcitabine + Cisplatin | Arm J: Nivolumab + Ipilimumab | Arm K: Nivolumab In Squamous Histology Subjects (NSCLC) | Arm L: Nivolumab In Non-squamous Histology Subjects (NSCLC) | Arm M: Nivolumab | Arm N: Nivolumab + Ipilimumab | Arm O: Nivolumab + Ipilimumab | Arm P: Nivolumab + Ipilimumab | Arm Q: Nivolumab + Ipilimumab | Arm B: Nivolumab + Pemetrexed + Cisplatin | Arm C: Nivolumab + Paclitaxel + Carboplatin | Arm D: Nivolumab + Bevacizumab Maintenance | Arm E: Nivolumab + Erlotinib | Arm F: Nivolumab | Arm G: Nivolumab + Ipilimumab | Arm H: Nivolumab + Ipilimumab | Arm I: Nivolumab + Ipilimumab
Serious Adverse Events (participants affected / at risk) | 4/12 | 12/16 | 3/13 | 4/13 | 4/12 | 12/31 | 21/40 | 25/38 | 25/39 | 10/15 | 17/29 | 3/12 | 11/21 | 23/52 | 6/9 | 12/15 | 5/9
Other Adverse Events (participants affected / at risk) | 12/12 | 16/16 | 11/13 | 13/13 | 11/12 | 30/31 | 33/40 | 35/38 | 33/39 | 15/15 | 29/29 | 11/12 | 21/21 | 50/52 | 9/9 | 15/15 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Nivolumab + Gemcitabine + Cisplatin (N=12) | Arm J: Nivolumab + Ipilimumab (N=16) | Arm K: Nivolumab In Squamous Histology Subjects (NSCLC) (N=13) | Arm L: Nivolumab In Non-squamous Histology Subjects (NSCLC) (N=13) | Arm M: Nivolumab (N=12) | Arm N: Nivolumab + Ipilimumab (N=31) | Arm O: Nivolumab + Ipilimumab (N=40) | Arm P: Nivolumab + Ipilimumab (N=38) | Arm Q: Nivolumab + Ipilimumab (N=39) | Arm B: Nivolumab + Pemetrexed + Cisplatin (N=15) | Arm C: Nivolumab + Paclitaxel + Carboplatin (N=29) | Arm D: Nivolumab + Bevacizumab Maintenance (N=12) | Arm E: Nivolumab + Erlotinib (N=21) | Arm F: Nivolumab (N=52) | Arm G: Nivolumab + Ipilimumab (N=9) | Arm H: Nivolumab + Ipilimumab (N=15) | Arm I: Nivolumab + Ipilimumab (N=9)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 1
Bandaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrioventricular block (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 3 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hypophysitis (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypopituitarism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Secondary adrenocortical insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blindness unilateral (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Uveitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vitreous haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 3 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Oesophageal fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tongue discolouration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bile duct stenosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Meningitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 3 | 1 | 2 | 1 | 1 | 1 | 0 | 1 | 1 | 2 | 2 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Radiation necrosis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 4 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Latent autoimmune diabetes in adults (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Embolic cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Facial nerve disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Miller fisher syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nervous system disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Vocal cord paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nephritis allergic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Renal salt-wasting syndrome (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 3 | 4 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 2 | 0 | 2 | 2 | 2 | 1 | 1 | 1 | 0 | 1 | 2 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 2 | 0 | 2 | 2 | 2 | 1 | 1 | 1 | 0 | 0 | 1 | 2 | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Aortic stenosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Superior vena cava syndrome (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Nivolumab + Gemcitabine + Cisplatin (N=12) | Arm J: Nivolumab + Ipilimumab (N=16) | Arm K: Nivolumab In Squamous Histology Subjects (NSCLC) (N=13) | Arm L: Nivolumab In Non-squamous Histology Subjects (NSCLC) (N=13) | Arm M: Nivolumab (N=12) | Arm N: Nivolumab + Ipilimumab (N=31) | Arm O: Nivolumab + Ipilimumab (N=40) | Arm P: Nivolumab + Ipilimumab (N=38) | Arm Q: Nivolumab + Ipilimumab (N=39) | Arm B: Nivolumab + Pemetrexed + Cisplatin (N=15) | Arm C: Nivolumab + Paclitaxel + Carboplatin (N=29) | Arm D: Nivolumab + Bevacizumab Maintenance (N=12) | Arm E: Nivolumab + Erlotinib (N=21) | Arm F: Nivolumab (N=52) | Arm G: Nivolumab + Ipilimumab (N=9) | Arm H: Nivolumab + Ipilimumab (N=15) | Arm I: Nivolumab + Ipilimumab (N=9)
Anaemia (Blood and lymphatic system disorders) | 8 | 1 | 1 | 0 | 0 | 4 | 5 | 6 | 5 | 2 | 8 | 0 | 0 | 2 | 1 | 1 | 2
Granulocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 1 | 0 | 0 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 0 | 0 | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 1 | 0 | 0 | 0 | 0
Polycythaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Deafness (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Deafness unilateral (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 5 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Autoimmune thyroiditis (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 2 | 0 | 0 | 1 | 2 | 2 | 2 | 4 | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 0
Hypophysitis (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 1 | 2 | 1 | 0 | 2 | 6 | 4 | 5 | 1 | 1 | 1 | 3 | 4 | 1 | 2 | 1
Thyroiditis (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Astigmatism (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Chalazion (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 2 | 2 | 1 | 1 | 1 | 0 | 0 | 0
Eye discharge (Eye disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Eye pruritus (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Eye swelling (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Eyelid oedema (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 2 | 2 | 5 | 0 | 2 | 1 | 0 | 1 | 0
Visual impairment (Eye disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 1 | 1
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 2 | 1 | 2 | 3 | 3 | 4 | 4 | 1 | 2 | 1 | 2 | 5 | 0 | 2 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 6 | 1 | 0 | 0 | 1 | 1 | 4 | 0 | 0 | 0
Anogenital dysplasia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 10 | 6 | 0 | 1 | 3 | 6 | 11 | 8 | 10 | 6 | 15 | 1 | 9 | 17 | 2 | 3 | 1
Defaecation urgency (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 6 | 5 | 1 | 1 | 11 | 13 | 10 | 12 | 5 | 14 | 2 | 10 | 15 | 4 | 10 | 2
Dry mouth (Gastrointestinal disorders) | 1 | 3 | 1 | 1 | 0 | 5 | 5 | 3 | 4 | 0 | 0 | 0 | 5 | 5 | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 4 | 2 | 3 | 2 | 2 | 0 | 1 | 1 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 2 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eructation (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 2
Gastric disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 3 | 2 | 2 | 2 | 1 | 2 | 0 | 1 | 0 | 1 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 8 | 8 | 2 | 0 | 2 | 9 | 12 | 10 | 11 | 12 | 12 | 3 | 10 | 17 | 2 | 6 | 3
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Periodontal disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sensitivity of teeth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Steatorrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 3 | 0 | 2 | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 7 | 0 | 0 | 2 | 2 | 8 | 5 | 5 | 6 | 9 | 1 | 7 | 7 | 2 | 2 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 2 | 2 | 0 | 1 | 1 | 1 | 1 | 0 | 0
Catheter site erythema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site pruritus (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 1 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Chest pain (General disorders) | 2 | 1 | 0 | 1 | 0 | 2 | 2 | 1 | 3 | 1 | 2 | 1 | 2 | 1 | 0 | 1 | 0
Chills (General disorders) | 1 | 2 | 2 | 0 | 1 | 3 | 1 | 5 | 5 | 1 | 1 | 1 | 1 | 2 | 1 | 4 | 0
Decreased activity (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Energy increased (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 10 | 11 | 6 | 7 | 7 | 16 | 13 | 14 | 18 | 14 | 23 | 6 | 16 | 28 | 4 | 11 | 6
Feeling cold (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 2 | 0 | 2 | 1 | 0 | 0 | 0
Gastrointestinal disorder (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Implant site oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 2 | 0 | 0 | 0 | 3 | 3 | 1 | 2 | 1 | 3 | 1 | 0 | 1 | 0 | 0 | 0
Infusion site irritation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site reaction (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 1 | 0
Mucosal inflammation (General disorders) | 2 | 2 | 0 | 0 | 1 | 2 | 1 | 1 | 1 | 1 | 5 | 2 | 2 | 1 | 0 | 0 | 0
Nodule (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 4 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Oedema peripheral (General disorders) | 1 | 0 | 0 | 3 | 1 | 4 | 2 | 7 | 1 | 2 | 5 | 2 | 2 | 2 | 2 | 0 | 0
Pain (General disorders) | 1 | 0 | 1 | 1 | 0 | 4 | 1 | 4 | 3 | 0 | 2 | 0 | 2 | 3 | 1 | 3 | 0
Peripheral swelling (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Pneumonia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 2 | 2 | 3 | 0 | 5 | 4 | 9 | 7 | 0 | 9 | 1 | 5 | 6 | 2 | 6 | 0
Temperature intolerance (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Xerosis (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 2 | 0 | 0 | 0
Autoimmune disorder (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 5 | 0 | 0 | 2 | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Alpha haemolytic streptococcal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Angular cheilitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Body tinea (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Candida infection (Infections and infestations) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Genital herpes (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes virus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0
Metapneumovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nail infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 1 | 1 | 1 | 1 | 2 | 2 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pilonidal cyst (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 3 | 3 | 2 | 0 | 1 | 3 | 2 | 0 | 3 | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 3 | 4 | 1 | 3 | 0 | 0 | 3 | 3 | 2 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 1 | 1 | 0 | 1 | 2 | 1 | 4 | 3 | 2 | 3 | 0 | 0 | 4 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Contrast media reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1 | 3 | 0 | 2 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 1 | 1 | 0 | 0 | 2 | 0 | 1 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 1 | 0 | 0 | 1 | 3 | 0 | 4 | 3 | 1 | 2 | 1 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Post procedural contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Procedural vomiting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Urinary retention postoperative (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 8 | 1 | 1 | 1 | 1 | 0 | 3 | 2 | 0 | 4 | 1
Amylase increased (Investigations) | 0 | 2 | 2 | 2 | 1 | 5 | 2 | 8 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 3 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 2 | 8 | 1 | 1 | 1 | 0 | 0 | 3 | 2 | 0 | 4 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood corticotrophin decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 3 | 0 | 0 | 2 | 0 | 5 | 3 | 1 | 3 | 0 | 1 | 0 | 0 | 2 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood potassium decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood thyroid stimulating hormone decreased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Breath sounds abnormal (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Creatinine renal clearance decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Csf protein increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 1
Heart rate increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 2 | 1 | 1 | 1 | 5 | 3 | 8 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 2
Lymphocyte count decreased (Investigations) | 1 | 0 | 1 | 0 | 0 | 1 | 4 | 3 | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 1
Thyroxine increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0
Tri-iodothyronine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Troponin t increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urine output decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 2 | 1 | 1 | 0 | 1 | 4 | 5 | 7 | 0 | 3 | 1 | 2 | 4 | 1 | 3 | 1
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 8 | 8 | 1 | 3 | 2 | 4 | 8 | 11 | 14 | 9 | 10 | 1 | 6 | 9 | 6 | 6 | 3
Dehydration (Metabolism and nutrition disorders) | 1 | 3 | 0 | 1 | 0 | 1 | 3 | 1 | 5 | 1 | 2 | 0 | 3 | 3 | 0 | 4 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 3 | 1 | 0 | 2 | 1 | 6 | 0 | 0 | 2 | 1 | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 3 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 3 | 2 | 1 | 2 | 0 | 2 | 1 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 3 | 0 | 0 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 2 | 3 | 2 | 3 | 0 | 1 | 1 | 0 | 1 | 1 | 2 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 3 | 1 | 1 | 2 | 9 | 11 | 8 | 4 | 5 | 14 | 3 | 4 | 9 | 1 | 4 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 4 | 1 | 4 | 0 | 1 | 3 | 3 | 11 | 3 | 7 | 1 | 7 | 8 | 1 | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | 0 | 1 | 2 | 0 | 3 | 0 | 3 | 1 | 3 | 4 | 1 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 4 | 2 | 3 | 1 | 1 | 1 | 2 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0 | 0 | 1 | 2 | 2 | 3 | 0 | 4 | 1 | 5 | 4 | 1 | 1 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 4 | 1 | 0 | 3 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 2 | 1 | 3 | 4 | 1 | 2 | 0 | 4 | 3 | 5 | 7 | 2 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 0 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1 | 1 | 2 | 5 | 5 | 4 | 5 | 1 | 8 | 0 | 4 | 5 | 0 | 1 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 0 | 2 | 2 | 4 | 5 | 1 | 1 | 2 | 1 | 0 | 1 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 1 | 4 | 3 | 3 | 7 | 0 | 5 | 3 | 4 | 8 | 0 | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Autonomic neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 2 | 1 | 1 | 2 | 1 | 4 | 3 | 2 | 3 | 3 | 3 | 3 | 7 | 0 | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 2 | 1 | 0 | 2 | 0 | 1 | 0 | 4 | 3 | 3 | 5 | 1 | 3 | 2 | 1 | 2 | 0
Headache (Nervous system disorders) | 1 | 3 | 1 | 1 | 0 | 5 | 5 | 6 | 6 | 3 | 9 | 1 | 4 | 3 | 0 | 3 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 2 | 1 | 1 | 0 | 2 | 1 | 1 | 1 | 5 | 0 | 1 | 1 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 14 | 3 | 1 | 4 | 0 | 2 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 1 | 2 | 1 | 0 | 0 | 1 | 2 | 6 | 1 | 0 | 0 | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tension headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 2 | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 3 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 1 | 0 | 1 | 0 | 2 | 2 | 2 | 4 | 0 | 1 | 0 | 1 | 3 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 0 | 0 | 1 | 6 | 4 | 7 | 6 | 2 | 6 | 0 | 1 | 9 | 0 | 1 | 1
Mental fatigue (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mood altered (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bladder pain (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Stress urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary straining (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Menopausal symptoms (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Penile haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 6 | 3 | 8 | 5 | 11 | 12 | 13 | 13 | 5 | 15 | 7 | 9 | 28 | 3 | 6 | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1 | 2 | 1 | 0 | 2 | 0 | 3 | 2 | 1 | 6 | 1 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 1 | 2 | 0 | 13 | 9 | 12 | 11 | 8 | 15 | 5 | 7 | 17 | 2 | 5 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 2 | 2 | 1 | 1 | 1 | 3 | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 5 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 2 | 0 | 2 | 1 | 3 | 2 | 4 | 1 | 1 | 0 | 2 | 2 | 0 | 1 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 1 | 4 | 0 | 1 | 0
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 5 | 5 | 1 | 3 | 0 | 3 | 5 | 0 | 1 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 3 | 2 | 3 | 0 | 3 | 5 | 0 | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 2 | 2 | 1 | 0 | 2 | 1 | 3 | 1 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0 | 1 | 2 | 1 | 2 | 1 | 1 | 2 | 0 | 1 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 3 | 2 | 3 | 1 | 4 | 3 | 5 | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 3 | 5 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 4 | 1 | 2 | 0 | 0 | 0
Vocal cord disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 3 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 2 | 15 | 0 | 3 | 1 | 1 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 1 | 3 | 4 | 2 | 6 | 3 | 0 | 2 | 5 | 5 | 0 | 1 | 0
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 3 | 2 | 1 | 0 | 0
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 1
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 2 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 4 | 1 | 0 | 0 | 8 | 5 | 16 | 7 | 2 | 3 | 1 | 5 | 15 | 2 | 4 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 6 | 3 | 1 | 1 | 11 | 14 | 8 | 6 | 6 | 10 | 2 | 13 | 15 | 2 | 6 | 2
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 4 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 3 | 1 | 0 | 0 | 4 | 4 | 7 | 4 | 1 | 1 | 1 | 1 | 1 | 1 | 2 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 1 | 4 | 0 | 2 | 0 | 1 | 2 | 1 | 0 | 1
Scab (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 5 | 1 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin hypertrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin plaque (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Solar dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arterial thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 2 | 1 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hot flush (Vascular disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 3 | 4 | 2 | 4 | 1 | 1 | 2 | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 4 | 1 | 2 | 1 | 2 | 1 | 0 | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vena cava thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.